CLINICAL TRIAL: NCT01927549
Title: Prospective Randomized Multicenter Study Comparing Immediate Multivessel Revascularization by PCI Versus Culprit Lesion PCI With Staged Non-culprit Lesion Revascularization in Patients With Acute Myocardial Infarction Complicated by Cardiogenic Shock
Brief Title: Culprit Lesion Only PCI Versus Multivessel PCI in Cardiogenic Shock
Acronym: CULPRIT-SHOCK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: European Commission (Other); German Cardiac Society (Other); Deutsche Stiftung für Herzforschung (Other); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Holger Thiele, Coordinator, Heart Center Leipzig - University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CULPRIT-SHOCK1.2
Record Dates: First submitted 2013-08-14; First posted 2013-08-22 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Cardiogenic Shock; Acute Myocardial Infarction; Complications
Keywords: cardiogenic shock; infarction; multivessel coronary artery disease; angioplasty
MeSH Terms: conditions — Shock, Cardiogenic; Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate multivessel PCI (Active Comparator): After diagnostic angiography the culprit lesion is identified and PCI should be performed using standard techniques. The use of drug-eluting stents is recommended but not mandatory. All additional lesions in other major coronary arteries defined by a diameter >2 mm with high grade stenoses (>70% by visual assessment) should be intervened using standard techniques. Other major coronary arteries are defined by stenoses of other vessels and are not confined to a diagonal branch if the left anterior descending coronary artery was identified as the culprit lesion.
  Interventions: Procedure: Immediate multivessel PCI
- Culprit lesion only PCI (Active Comparator): After diagnostic angiography the culprit lesion is identified and PCI of the culprit lesion should be performed using standard techniques. The use of drug-eluting stents is recommended but not mandatory. All other lesions should be left untreated in the acute setting. Complete revascularization of the non-culprit lesions may be performed at a later time point as staged procedure depending on remaining ischemia (as per guideline recommendations either by PCI or CABG).
  Interventions: Procedure: Culprit Lesion only PCI

INTERVENTIONS:
Procedure: Immediate multivessel PCI
  Arms: Immediate multivessel PCI
Procedure: Culprit Lesion only PCI
  Arms: Culprit lesion only PCI

SUMMARY:
The study compares the therapies of instant multivessel balloon angioplasty plus stent implantation or the balloon angioplasty plus stent implantation of the infarct artery alone with any possible graduated later treatment of the other vessels in patients with acute myocardial infarction with cardioganic shock.

The main study hypothesis is to explore if culprit vessel only PCI with potentially subsequent staged revascularization in comparison to immediate multivessel revascularization by PCI in patients with cardiogenic shock complicating acute myocardial infarction reduces the incidence of 30- day mortality and/or severe renal failure requiring renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

Cardiogenic shock complicating acute myocardial infarction (STEMI or NSTEMI) with obligatory:

I) Planned early revascularization by PCI II) Multivessel coronary artery disease defined as more than 70% stenosis in at least 2 major vessels (more than 2 mm diameter) with identifiable culprit lesion III)

1. Systolic blood pressure less than 90 mmHg for more than 30 min or
2. catecholamines required to maintain pressure more than 90 mmHg during systole and IV) Signs of pulmonary congestion V) Signs of impaired organ perfusion with at least one of the following criteria

a) Altered mental status b) Cold, clammy skin and extremities c) Oliguria with urine output less than 30 ml/h d) Serum-lactate more than 2.0 mmol/l VI) Informed consent

Exclusion Criteria:

* Resuscitation more than 30 minutes
* No intrinsic heart action
* Cerebral deficit with fixed dilated pupils (not drug-induced)
* Need for primary urgent bypass surgery (to be determined after diagnostic angiography)
* Single vessel disease
* Mechanical cause of cardiogenic shock
* Onset of shock more than 12 h
* Massive lung emboli
* Age more than 90 years
* Shock of other cause (bradycardia, sepsis, hypovolemia, etc.)
* Other severe concomitant disease with limited life expectancy <6 months
* Pregnancy
* Known severe renal insufficiency (creatinine clearance <30 ml/kg)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2013-04; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
30-day mortality and/or severe renal failure requiring renal replacement therapy | 30 days

SECONDARY OUTCOMES:
30-day mortality | 30 days
Requirement of renal replacement therapy | 30 days
Time to hemodynamic stabilization | 30 days
Duration of catecholamine therapy | 30 days
Serial creatinine-level creatinine-clearance | 30 days
Length of ICU-stay | 30 days
Serial intensive care scoring (SAPS-II score) until stabilization | 30 days
Requirement and length of mechanical ventilation | 30 days
All-cause death within 12 months follow-up | 12 months
Recurrent infarction within 30-days follow-up | 30 days
Death or recurrent infarction at 12 months follow-up | 12 months
Rehospitalization for congestive heart failure within 12 months follow-up | 12 months
Death/recurrent infarction/rehospitalization for congestive heart failure within 12 months | 12 months
Need for repeat revascularization (PCI and/or CABG) within 12 months follow-up | 12 months
Peak creatine kinase level during hospital stay | 30 days
Quality of life at 6 and 12 months assessed using Euroqol 5D (EQ-5D) | 12 months
Maximum creatine kinase-MB level | 30 days
Maximum troponin level | 30 days
Recurrent infarction within 12 months follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Study Chair — Heart Center Leipzig - University Hospital
Locations (3):
- Germany (3):
  - University of Goettingen, Göttingen
  - Heart Center Leipzig - University Hospital, Leipzig
  - University of Leipzig - Heart Center, Leipzig

REFERENCES:
- [Derived] Jung C, Lang A, Duse DA, Bruno RR, Poss J, Wolff G, Ceglarek U, Zeymer U, Fuernau G, Zweck E, Desch S, Freund A, Isermann B, Pfeiler S, Wernly B, Kelm M, Thiele H, Gerdes N. Plasma Proteome Analysis Identifies Vascular Endothelial Growth Factor Receptor 1 as a Prognostic Biomarker in Cardiogenic Shock. Circ Heart Fail. 2025 Dec;18(12):e012890. doi: 10.1161/CIRCHEARTFAILURE.125.012890. Epub 2025 Oct 1. PMID 41031405
- [Derived] Zeymer-von Metnitz D, Ouarrak T, Huber K, Noc M, Desch S, Freund A, Zeymer U, Thiele H, Poss J. Mild Induced Hypothermia in Patients with Infarct-Related Cardiogenic Shock and Cardiac Arrest: Insights from the CULPRIT-SHOCK Trial. Eur Heart J Acute Cardiovasc Care. 2025 Sep 23:zuaf124. doi: 10.1093/ehjacc/zuaf124. Online ahead of print. PMID 40986817
- [Derived] Zeymer U, Alushi B, Noc M, Mamas MA, Montalescot G, Fuernau G, Huber K, Poess J, de Waha-Thiele S, Schneider S, Ouarrak T, Desch S, Lauten A, Thiele H. Influence of Culprit Lesion Intervention on Outcomes in Infarct-Related Cardiogenic Shock With Cardiac Arrest. J Am Coll Cardiol. 2023 Mar 28;81(12):1165-1176. doi: 10.1016/j.jacc.2023.01.029. PMID 36948733
- [Derived] Bohme M, Desch S, Rosolowski M, Scholz M, Krohn K, Buttner P, Cross M, Kirchberg J, Rommel KP, Poss J, Freund A, Baber R, Isermann B, Ceglarek U, Metzeler KH, Platzbecker U, Thiele H. Impact of Clonal Hematopoiesis in Patients With Cardiogenic Shock Complicating Acute Myocardial Infarction. J Am Coll Cardiol. 2022 Oct 18;80(16):1545-1556. doi: 10.1016/j.jacc.2022.08.740. PMID 36229091
- [Derived] Ceglarek U, Schellong P, Rosolowski M, Scholz M, Willenberg A, Kratzsch J, Zeymer U, Fuernau G, de Waha-Thiele S, Buttner P, Jobs A, Freund A, Desch S, Feistritzer HJ, Isermann B, Thiery J, Poss J, Thiele H. The novel cystatin C, lactate, interleukin-6, and N-terminal pro-B-type natriuretic peptide (CLIP)-based mortality risk score in cardiogenic shock after acute myocardial infarction. Eur Heart J. 2021 Jun 21;42(24):2344-2352. doi: 10.1093/eurheartj/ehab110. PMID 33647946
- [Derived] Hauguel-Moreau M, Barthelemy O, Farhan S, Huber K, Rouanet S, Zeitouni M, Guedeney P, Hage G, Vicaut E, Zeymer U, Desch S, Thiele H, Montalescot G. Culprit lesion location and outcomes in patients with multivessel disease and infarct-related cardiogenic shock: a core laboratory analysis of the CULPRIT-SHOCK trial. EuroIntervention. 2021 Aug 6;17(5):e418-e424. doi: 10.4244/EIJ-D-20-00561. PMID 32894227
- [Derived] Sag CM, Zeymer U, Ouarrak T, Schneider S, Montalescot G, Huber K, Fuernau G, Freund A, Feistritzer HJ, Desch S, Thiele H, Maier LS. Effects of ON-Hours Versus OFF-Hours Admission on Outcome in Patients With Myocardial Infarction and Cardiogenic Shock: Results From the CULPRIT-SHOCK Trial. Circ Cardiovasc Interv. 2020 Sep;13(9):e009562. doi: 10.1161/CIRCINTERVENTIONS.120.009562. Epub 2020 Sep 4. PMID 32883104
- [Derived] Farhan S, Vogel B, Montalescot G, Barthelemy O, Zeymer U, Desch S, de Waha-Thiele S, Maier LS, Sandri M, Akin I, Fuernau G, Ouarrak T, Hauguel-Moreau M, Schneider S, Thiele H, Huber K. Association of Culprit Lesion Location With Outcomes of Culprit-Lesion-Only vs Immediate Multivessel Percutaneous Coronary Intervention in Cardiogenic Shock: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2020 Dec 1;5(12):1329-1337. doi: 10.1001/jamacardio.2020.3377. PMID 32845312
- [Derived] Rubini Gimenez M, Zeymer U, Desch S, de Waha-Thiele S, Ouarrak T, Poess J, Meyer-Saraei R, Schneider S, Fuernau G, Stepinska J, Huber K, Windecker S, Montalescot G, Savonitto S, Jeger RV, Thiele H. Sex-Specific Management in Patients With Acute Myocardial Infarction and Cardiogenic Shock: A Substudy of the CULPRIT-SHOCK Trial. Circ Cardiovasc Interv. 2020 Mar;13(3):e008537. doi: 10.1161/CIRCINTERVENTIONS.119.008537. Epub 2020 Mar 10. PMID 32151161
- [Derived] Feistritzer HJ, Desch S, Zeymer U, Fuernau G, de Waha-Thiele S, Dudek D, Huber K, Stepinska J, Schneider S, Ouarrak T, Thiele H. Prognostic Impact of Atrial Fibrillation in Acute Myocardial Infarction and Cardiogenic Shock. Circ Cardiovasc Interv. 2019 Jun;12(6):e007661. doi: 10.1161/CIRCINTERVENTIONS.118.007661. Epub 2019 Jun 6. PMID 31167601
- [Derived] Thiele H, Akin I, Sandri M, de Waha-Thiele S, Meyer-Saraei R, Fuernau G, Eitel I, Nordbeck P, Geisler T, Landmesser U, Skurk C, Fach A, Jobs A, Lapp H, Piek JJ, Noc M, Goslar T, Felix SB, Maier LS, Stepinska J, Oldroyd K, Serpytis P, Montalescot G, Barthelemy O, Huber K, Windecker S, Hunziker L, Savonitto S, Torremante P, Vrints C, Schneider S, Zeymer U, Desch S; CULPRIT-SHOCK Investigators. One-Year Outcomes after PCI Strategies in Cardiogenic Shock. N Engl J Med. 2018 Nov 1;379(18):1699-1710. doi: 10.1056/NEJMoa1808788. Epub 2018 Aug 25. PMID 30145971
- [Derived] Thiele H, Akin I, Sandri M, Fuernau G, de Waha S, Meyer-Saraei R, Nordbeck P, Geisler T, Landmesser U, Skurk C, Fach A, Lapp H, Piek JJ, Noc M, Goslar T, Felix SB, Maier LS, Stepinska J, Oldroyd K, Serpytis P, Montalescot G, Barthelemy O, Huber K, Windecker S, Savonitto S, Torremante P, Vrints C, Schneider S, Desch S, Zeymer U; CULPRIT-SHOCK Investigators. PCI Strategies in Patients with Acute Myocardial Infarction and Cardiogenic Shock. N Engl J Med. 2017 Dec 21;377(25):2419-2432. doi: 10.1056/NEJMoa1710261. Epub 2017 Oct 30. PMID 29083953
- [Derived] Quayyum Z, Briggs A, Robles-Zurita J, Oldroyd K, Zeymer U, Desch S, Waha S, Thiele H. Protocol for an economic evaluation of the randomised controlled trial of culprit lesion only PCI versus immediate multivessel PCI in acute myocardial infarction complicated by cardiogenic shock: CULPRIT-SHOCK trial. BMJ Open. 2017 Aug 18;7(8):e014849. doi: 10.1136/bmjopen-2016-014849. PMID 28821512
- [Derived] Thiele H, Desch S, Piek JJ, Stepinska J, Oldroyd K, Serpytis P, Montalescot G, Noc M, Huber K, Fuernau G, de Waha S, Meyer-Saraei R, Schneider S, Windecker S, Savonitto S, Briggs A, Torremante P, Vrints C, Schuler G, Ceglarek U, Thiery J, Zeymer U; CULPRIT-SHOCK Investigators. Multivessel versus culprit lesion only percutaneous revascularization plus potential staged revascularization in patients with acute myocardial infarction complicated by cardiogenic shock: Design and rationale of CULPRIT-SHOCK trial. Am Heart J. 2016 Feb;172:160-9. doi: 10.1016/j.ahj.2015.11.006. Epub 2015 Dec 1. PMID 26856228
- [Derived] AbouEzzeddine OF, Lala A, Khazanie PP, Shah R, Ho JE, Chen HH, Pang PS, McNulty SE, Anstrom KJ, Hernandez AF, Redfield MM; NHLBI Heart Failure Clinical Research Network. Evaluation of a provocative dyspnea severity score in acute heart failure. Am Heart J. 2016 Feb;172:34-41. doi: 10.1016/j.ahj.2015.10.009. Epub 2015 Oct 20. PMID 26856213